CLINICAL TRIAL: NCT02330666
Title: Parent-child Communication and Health-risk Behavior
Acronym: MP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Loyola University Chicago (Other); Iowa State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2003-352
Record Dates: First submitted 2014-12-30; First posted 2015-01-05 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Parent-Child Relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comparison (No Intervention): Standard care
- Intervention (Experimental): Communication skills training Mission Possible: Parents & Kids Who Listen
  Interventions: Behavioral: Mission Possible: Parents & Kids Who Listen

INTERVENTIONS:
Behavioral: Mission Possible: Parents & Kids Who Listen — MP is a 12-hour, 6-session, manualized skills training program with 2 boosters. Behavioral strategies teach adults and youth to communicate with one another emphasizing youth's need for flexible family boundaries, emotional closeness, and adults as resources. Dyads attend together. Sessions begin with relaxation exercises, review of the prior week's lessons and homework, and examination of success and failure in trying communication techniques. New concepts are introduced using didactic videotaped presentations. Lively, interactive, developmentally appropriate group exercises follow reflective of ethnic diversity that are reinforced with handouts and encouragement to try them at home. Week-by-week content covers: Developmental Changes; Self-Esteem; Communicating What You Want; Listening to What the Other Wants; Solving Conflicts; and Letting Go. The booster sessions are 2 hours in length and update developmental concepts; 5 basic listening skills; and 6 conflict resolution steps.
  Arms: Intervention

SUMMARY:
Engaging in health-risk behaviors such as tobacco and alcohol use put youth at risk for health problems that may compromise their futures and are extremely costly to society. Positive parent-child communication, characterized by openness, satisfaction with the family, caring, and effective problem-solving, has been found to be protective against a youth's involvement in health-risk behaviors. To promote positive adult-youth communication, in earlier work we developed, tested, and found efficacious an intervention, Mission Possible: Parents and Kids Who Listen (MP). This study is designed to test the following hypotheses: (a) Adults and youth who participate in MP will demonstrate more positive communication when compared with adults who did not participate; (b) Youth who participate in MP will have a lower incidence of health-risk behavior when compared with youth who did not participate; and (c) Positive adult-youth communication will mediate childhood health-risk behavior in the presence of risk processes that predict participation. The experimental design is a 2-group (intervention and comparison) pre-test repeated measures design with six waves of data collection over three years and two booster sessions of the intervention. Elementary school and community centers in Madison and Chicago served as recruitment sites for parent-child dyads.

ELIGIBILITY:
Inclusion Criteria:

* Adults and youth must be English speakers
* Youth must be 10 years old

Exclusion Criteria:

* Severe mental or physical illness that could preclude involvement in data collection procedures
* Family plans to move from the metropolitan areas prior to study completion

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2004-08; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Youth Health Risk Behavior | 3 years
  Measured with the 22-item Children's Health Risk Behavior Scale (CHRBS). This instrument, based on the conceptual categories of the Youth Risk Behavioral Surveillance Survey, assesses potential for unintentional and intentional injury or violence, tobacco use, alcohol and other drug use, sexual curiosity, and health practices.

SECONDARY OUTCOMES:
Openness of Communication | 3 years
  The Parent Adolescent Communication Inventory (Olson, 1983) is a 20-item, 2-subscale (open or problem communication) self-report instrument with a youth version and an adult version, the difference being the target of the item - mother/father or youth. Scores are computed for adult communication, youth-mother communication, youth-father communication.
Family Satisfaction | 3 years
  The Family Adaptability and Cohesion Evaluation Scale III is a 20-item, self-report instrument (Olson, 1994) to measure family satisfaction. Participants answer the items twice, first to assess current and then to assess ideal family system conditions. The difference between ideal and perceived conditions yields a family satisfaction score.
Problem-Solving Skill | 3 years
  50% of the dyads were randomly selected for assessment of problem solving ability. The procedure was to (a) identify a problem for discussion from the Issues Checklist (IC), (b) videotape the dyad attempting to solve the problem identified, and (c) code the videotaped interaction using the Iowa Family Interaction Rating Scales (IFIRS). The IFIRS is a macro-level observational coding system that was initially developed in 1989 and has undergone 5 revisions. Scales used to assess three aspects of family interaction were: (a) individual behavioral characteristics or each person's generalized interaction consisting of 8 items, e.g., use of humor, mood, whining and complaining; (b) dyadic behavioral characteristics or the nature of behavior exchanged from one family member to another consisting of 22 items, e.g., hostility, warmth/support; and (c) the family problem-solving process consisting of 10 items, e.g., solution quality, family enjoyment.

CONTACTS AND LOCATIONS:
Overall Officials: Susan K Riesch, PhD, Principal Investigator — University of Wisconsin, Madison